CLINICAL TRIAL: NCT05857137
Title: Investigational TMS Study of Cognitive Impairment in Early Psychosis
Brief Title: Psychosis TMS Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hamdi Eryilmaz, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2018P000014
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Psychosis
Keywords: Cognitive impairment; Transcranial Magnetic Stimulation; Attention; Short-term memory
MeSH Terms: conditions — Psychotic Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): Participants will receive single-session administration of TMS. Functional MRI will be acquired before and immediately after the intervention.
  Interventions: Device: Active TMS
- Placebo TMS (Placebo Comparator): Participants will also receive single session administration of placebo TMS (at least two days apart from the day of the active TMS). Functional MRI will be acquired before and immediately after the intervention.
  Interventions: Device: Placebo TMS

INTERVENTIONS:
Device: Active TMS — Continuous theta burst stimulation (cTBS) will be administered over the left inferior parietal lobule for approximately 3 minutes at 120% of the resting motor threshold.
  Arms: Active TMS
Device: Placebo TMS — Placebo TMS will be applied over the left inferior parietal lobule for approximately 3 minutes.
  Arms: Placebo TMS

SUMMARY:
The main goal of this study is to investigate the neural mechanisms of working memory function in patients with early psychosis using Transcranial Magnetic Stimulation (TMS) in conjunction with functional MRI. TMS is a noninvasive method used to modulate brain activity via changing magnetic fields applied over the surface of the scalp.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psychosis, psychosis not otherwise specified, schizophrenia, schizoaffective disorder, delusional disorder, bipolar disorder with psychosis, and schizophreniform disorder within first ten years of onset of psychotic symptoms.
* Ability to provide informed consent

Exclusion Criteria:

* TMS incompatibility including metallic implants in head and neck, cardiac pacemakers, history of seizures, pregnancy.
* MRI-incompatibility including implanted aneurism clips, cardiac pacemakers, metal implants, intrauterine devices, tattoos containing metal ink, pregnancy, and claustrophobia
* Severe substance abuse within 3 months (nicotine allowed)
* Unstable medical or neurologic illness that would preclude participation in study procedures

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Working memory accuracy | 2 hours
  Accuracy at high memory loads during performance of the Sternberg Item Recognition Paradigm will be assessed before and after the TMS interventions.
Reaction time during working memory | 2 hours
  Reaction time during performance of the Sternberg Item Recognition Paradigm will be assessed before and after the TMS interventions.
Resting state functional connectivity between the left inferior parietal lobule and the regions of the frontoparietal control network | 2 hours
  Functional connectivity between left inferior parietal lobule and dorsolateral prefrontal cortex will be computed during resting state acquired before and after the TMS interventions.
Resting state functional connectivity within the default mode network | 2 hours
  Functional connectivity between left inferior parietal lobule and other regions of the default mode network (including the posterior cingulate cortex and the medial prefrontal cortex) will be computed during resting state acquired before and after the TMS interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No